CLINICAL TRIAL: NCT01030900
Title: Phase II Trial of Alemtuzumab (Campath) and Dose-Adjusted EPOCH-Rituximab (DA-EPOCH-R) in Relapsed or Refractory Diffuse Large B-Cell and Hodgkin Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Wyndham Wilson, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100011; 10-C-0011
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Hodgkin Lymphoma; Diffuse Large B-Cell Lymphoma
Keywords: Immunosuppression; Microenvironment; Hodgkin Lymphoma; Microarray; B-Cell Lymphoma; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — Alemtuzumab; Rituximab; Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath (Experimental): Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin (EPOCH) + Rituximab + campath every 3 weeks for six cycles
  Interventions: Biological: Campath; Biological: Rituximab; Drug: EPOCH

INTERVENTIONS:
Biological: Campath — campath plus etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) and rituximab every 3 weeks for up to 6 cycles
  Other Names: Alemtuzumab
Biological: Rituximab — rituximab plus etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) and campath every 3 weeks for up to 6 cycles
  Other Names: Rituxan
Drug: EPOCH — Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) plus rituximab and campath every 3 weeks for up to 6 cycles
  Other Names: Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin

SUMMARY:
Background:

* Studies conducted at the National Cancer Institute suggest that certain chemotherapy drugs may be more effective if given by continuous infusion into the vein rather than by the standard method of rapid intravenous injection. One combination of six chemotherapy drugs, known as etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R), has had a high degree of effectiveness in people with certain kinds of cancer.
* Recent evidence also indicates that the effects of chemotherapy may be improved by combining the treatment with monoclonal antibodies, which are purified proteins that are specially made to attach to foreign substances such as cancer cells. A monoclonal antibody called campath (alemtuzumab) has been manufactured to attach to a protein called Campath-1 antigen (CD52) that may target tumor cells or the surrounding inflammatory cells.
* Researchers are interested in developing new treatments for large B-cell lymphoma or Hodgkin lymphoma that can best be treated with chemotherapy. This protocol is specifically for people with diffuse large B-cell or Hodgkin lymphomas that have not responded to standard treatments.

Objectives:

- To test whether giving campath (alemtuzumab) in combination with continuous infusion EPOCH-R chemotherapy will improve the outcome of lymphoma treatment.

Eligibility:

- Individuals 18 years of age and older who have large B-cell lymphoma or Hodgkin lymphoma that has not responded well to standard treatments.

Design:

* During the study, patients will receive standard EPOCH-R chemotherapy, which includes the following drugs: etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab. The additional drug, campath, will be given by intravenous (IV) infusion on the first day of treatment over several hours.
* When the campath IV infusion and rituximab IV infusion are complete, the drugs doxorubicin, etoposide, and vincristine will each be given by continuous IV infusion over the next 4 days (that is, continuously for a total of 96 hours). Cyclophosphamide will be given by IV infusion over several hours on Day 5. Prednisone will be given by mouth twice each day for 5 days.
* Patients may be given other drugs to treat the side effects of chemotherapy, to prevent possible infections, and to improve white blood cell counts.
* The campath-EPOCH-R therapy will be repeated every 21 days, as a cycle of therapy, for a total of 6 cycles. Following the fourth and sixth treatment cycles (approximately weeks 12 and 18) of campath-EPOCH-R treatment, study researchers will perform blood tests and computed tomography (CT)/magnetic resonance imaging (MRI) scans on all patients to assess their response to the treatment.

DETAILED DESCRIPTION:
Background:

Two signatures of the microenvironment were recently identified that are predictive of outcome in patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL), treated with rituximab, cyclophosphamide, hydroxydaunorubicin hydrochloride (doxorubicin hydrochloride), vincristine (Oncovin) and prednisone (R-CHOP). These signatures, called stromal 1 and stromal 2, are associated with genes expressed by infiltrating mononuclear cells. The stromal 2 signature, which includes genes associated with angiogenesis, is predictive of an inferior outcome. Based on these observations, we are interested in targeting the reactive cells in the microenvironment as a therapeutic strategy in patients with relapsed and refractory DLBCL. Along the same principles, we are also including patients with relapsed Hodgkin lymphoma (HL). The surrounding reactive cells around Hodgkin Reed Sternberg (HRS) cells are now not thought to be bystander cells and they appear to provide important survival signals to HRS cells.

* Campath-1 antigen (CD52) is one such promising target that is highly expressed in most of these infiltrating cells and on most DLBCL although not on HRS cells specifically. Anti-CD52 antibodies may have therapeutic value by depleting reactive B and T cells, and monocytes from the microenvironment.
* The dose of alemtuzumab in combination with dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH) is 30 mg intravenous (IV), as determined by a prior study done in patients with untreated peripheral T-cell lymphoma. The main toxicities of this combination are myelosuppression and opportunistic infections.
* An important component of this study will be to obtain tumor tissue for gene expression profiling and to assess microenvironment signatures and look at other molecular signatures and targets before treatment and in patients who progress and ultimately correlate response and outcome with these various end-points.

Objectives:

- Assess response, progression free survival (PFS) and overall survival (OS) in relapsed/refractory DLBCL and Hodgkin Lymphoma.

Eligibility:

* Previously treated or refractory classical large B-cell lymphomas, Grey-zone lymphoma and Hodgkin lymphoma, including Lymphocyte predominant Hodgkin Lymphoma (LPHL).
* Age greater than or equal to 18 years with adequate organ functions.
* Human immunodeficiency virus (HIV) negative and no active central nervous system (CNS) lymphoma.

Study Design:

* Patients will receive 30mg of Alemtuzumab on day 1 of therapy, followed by Rituximab on day 1 and dose-adjusted EPOCH chemotherapy days 1-5, up to six cycles of therapy.
* Tumor biopsies will be done before treatment, after 1 cycle of therapy and at relapse.
* It is anticipated that up to 10-15 patients per year may be enrolled onto this trial. Thus, accrual of up to 52 patients is expected to require approximately 4-5 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Previously treated or refractory classical large B-cell lymphomas, Grey-zone lymphoma and Hodgkin lymphoma, including Lymphocyte predominant Hodgkin Lymphoma (LPHL).
  2. Confirmed pathological diagnosis by the Laboratory of Pathology, National Cancer Institute (NCI).
  3. Age greater than or equal to 18 years.
  4. Eastern Cooperative Oncology Group (ECOG) performance 0-2
  5. Laboratory tests: absolute neutrophil count (ANC) greater than or equal to 1000/mm(3), platelet greater than or equal to 75,000/mm(3). Creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than or equal to 60 ml/min; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 5 times the upper limit of normal (ULN). Total bilirubin < 2.0 mg/dl except < 5mg/dL in patients with Gilbert's (as defined as > 80% unconjugated hyperbilirubinemia without other known cause); unless impairment due to organ involvement by lymphoma.

EXCLUSION CRITERIA:

1. Active symptomatic ischemic heart disease, myocardial infarction or congestive heart failure within the past year. If echocardiogram (ECHO) is obtained, the left ventricular ejection fraction (LVEF) should exceed 40%.
2. Human immunodeficiency virus (HIV) positive, because of the unknown effects of combined therapy with chemotherapy and an immunosuppressive agent on HIV progression.
3. Female subject of child-bearing potential not willing to use an acceptable method of birth control (i.e. a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and two years beyond treatment completion.
4. Female subject pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotrophin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for women without childbearing potential.
5. Male subject unwilling to use an acceptable method for contraception for the duration of the study and one year beyond treatment completion.
6. Invasive or active malignancy in past 2 years.
7. Serious concomitant medical illnesses that would jeopardize the patient s ability to receive the regimen with reasonable safety.
8. Active central nervous system (CNS) lymphoma. These patients have a poor prognosis and because they frequently develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events.
9. Systemic cytotoxic therapy within 3 weeks of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10-22 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H Wilson, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0011.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath: Participants will receive 30mg of Alemtuzumab on day 1 of therapy, followed by Rituximab on day 1 and dose-adjusted EPOCH chemotherapy days 1-5, up to six cycles of therapy.
Period: Overall Study
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
Started | 50
Completed | 48
Not Completed | 2
Not completed — Not treated due to congestive heart failure | 1
Not completed — Not treated due to rapid disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 44
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 43 [18 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 37
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50
Histology [Count of Participants; unit: Participants] — Grey Zone: cancer of a part of the immune system. Hodgkin lymphoma: cancer of the lymphatic system. Primary mediastinal B-cell lymphoma: cancer of the mature B-lymphocytes. Diffuse large B-cell lymphoma: cancer in the lymphocytes. T-cell histiocyte rich diffuse: malignancy of B-cells.
  Participants
    Grey-Zone | 4
    Hodgkin Lymphoma | 16
    Primary mediastinal B-cell lymphoma (PMBL) | 5
    Diffuse large B-cell lymphoma (DLBCL) | 23
    B-cell lymphoma not otherwise specified (NOS) | 2
Median Number of Prior Lines of Therapy [Median (Full Range); unit: lines of therapy] — Previous treatments received that were followed by disease assessment for the same diagnosis prior to enrolling on this study.
  lines of therapy | 2 [1 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is the time interval from start of treatment to documented evidence of disease progression estimated using a Kaplan Meier curve. Progression was assessed by the International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphomas and is defined as ≥50% increase from nadir in the sum of the products of diameters of any previously identified abnormal node for partial response or non-responders. And an appearance of any new lesion during or at the end of therapy.
Time Frame: Time of progression or death, approximately 10 months
Population: 48/50 participants were evaluable for this outcome measure because 2 participants were not treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
Number analyzed (Participants) | 48
months | 6.6 [3.3 to 8.8]

2. Primary Outcome: Overall Survival (OS)
Description: OS is from enrollment to the day of death estimated using the Kaplan-Meier curve.
Time Frame: Median overall survival from enrollment to the day of death, approximately 17.9 months
Population: 48/50 participants were evaluable for this outcome measure because 2 participants were not treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
Number analyzed (Participants) | 48
months | 17.9 [11.5 to 49.6]

3. Secondary Outcome: Clinical Response on Study and at Relapse After Dose Adjusted - Etoposide + Prednisone + Vincristine + Cyclophosphamide + Doxorubicin + Rituximab (DA-EPOCH-RC)
Description: Clinical response was assessed by the International Workshop to Standardize Response Criteria for non-Hodgkin's Lymphomas. Complete remission is complete disappearance of all detectable clinical and radiographic evidence of disease. Complete response unconfirmed is as per complete remission except that if a residual node is greater than 1.5cm, it must have decreased by greater than 75% in the sum of the products of the perpendicular diameters (SPD). Partial response is ≥50% decreased in the SPD of 6 largest dominant nodes or nodal masses. Relapsed disease is appearance of any new lesion or increase by ≥50% in the size of the previously involved sites. Stable disease is defined as less than a partial response but not progressive disease. Progression is ≥50% increase from nadir in the SPD of diameters of any previously identified abnormal node for partial response or non-responders; and an appearance of any new lesion during or at the end of therapy.
Time Frame: On study and at relapse after study treatment, approximately 10 months
Population: 46/50 participants were evaluable for this outcome measure because 2 participants were not treated, and two participants were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
Number analyzed (Participants) | 46
Participants
  Complete remission | 17
  Complete response unconfirmed | 0
  Partial response | 13
  Stable disease | 2
  Relapsed disease | 0
  Progressive disease | 14

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 58 months and 18 days.
Population: 2/50 participants were not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
Number analyzed (Participants) | 48
Participants | 48

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 58 months and 18 days.
Description: 2/50 participants were not treated.
Arm/Group | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath
All-Cause Mortality (participants affected / at risk) | 30/48
Serious Adverse Events (participants affected / at risk) | 27/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath (N=48)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 (36)
Fever (General disorders) | 4 (4)
Hypotension (Vascular disorders) | 2 (2)
Infections and infestations - Other, E.coli (Infections and infestations) | 1 (1)
Infections and infestations - Other, pseudomonas (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin + Rituximab + Campath (N=48)
Abdominal pain (Gastrointestinal disorders) | 5 (8)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (20)
Alkaline phosphatase increased (Investigations) | 4 (6)
Allergic reaction (Immune system disorders) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17)
Anal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 43 (130)
Anorectal infection (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Anxiety (Psychiatric disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 11 (16)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bladder infection (Infections and infestations) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Blood and lymphatic system disorders - Other, Amylase Ser (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (4)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (19)
Cluster of differentiation 4 (CD4) lymphocytes decreased (Investigations) | 12 (13)
Creatine phosphokinase (CPK) increased (Investigations) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 10 (12)
Cardiac disorders - Other, orthostasis (Cardiac disorders) | 1 (1)
Cardiac troponin I increased (Cardiac disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 18 (23)
Constipation (Gastrointestinal disorders) | 18 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Creatinine increased (Investigations) | 4 (5)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 7 (8)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 18 (26)
Dizziness (Nervous system disorders) | 9 (12)
Dry eye (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 5 (5)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 24 (27)
Febrile neutropenia (Blood and lymphatic system disorders) | 20 (37)
Fever (General disorders) | 19 (21)
Flu like symptoms (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 15 (20)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 31 (48)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 10 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (12)
Hyponatremia (Metabolism and nutrition disorders) | 8 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 17 (29)
Hypotension (Vascular disorders) | 9 (12)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, C. Diff (Infections and infestations) | 2 (2)
Infections and infestations - Other, cytomegalovirus (CMV) (Infections and infestations) | 4 (4)
Infections and infestations - Other, herpes simplex virus (HSV) (Infections and infestations) | 1 (1)
Infections and infestations - Other, Klebsiella pan S (Infections and infestations) | 1 (1)
Infections and infestations - Other, Wound (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Lymphocyte count decreased (Investigations) | 45 (120)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 21 (32)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (30)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - Other, Autonomic Neuropathy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, recurrent laryngeal nerve palsy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, sensory (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 43 (137)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (17)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (22)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 44 (140)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 2 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal mucositis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (3)
Sepsis (Infections and infestations) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Thromboembolic event (Vascular disorders) | 10 (10)
Tinnitus (Ear and labyrinth disorders) | 1 (2)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 8 (10)
Urinary tract pain (Renal and urinary disorders) | 4 (4)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 10 (13)
Watering eyes (Eye disorders) | 2 (2)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 47 (167)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT01030900/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT01030900/ICF_001.pdf